CLINICAL TRIAL: NCT00769470
Title: A Multicenter, Open Label, Randomized Phase II Trial of Presurgical Treatment With Single-Agent Trastuzumab (H) or Lapatinib (Ty) or the Combination of Trastuzumab and Lapatinib (H+Ty), Followed by Six Cycles of Docetaxel (T) and Carboplatin (C) With Trastuzumab (TCH) or Lapatinib (TCTy) or the Combination of Trastuzumab and Lapatinib (TCHTy) in Patients With HER2/Neu-Amplified Operable Breast Cancer
Brief Title: Docetaxel, Carboplatin, and Trastuzumab and/or Lapatinib in Treating Women With Stage I, Stage II, or Stage III Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000616008; P30CA016042 (NIH); TRIO-TORI-B-07; SANOFI-AVENTIS-TRIO-TORI-B-07; WIRB-20080822; NCT02668939 (obsolete NCT alias)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Docetaxel; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Active Comparator): Patients receive trastuzumab IV over 90 minutes on day in course 1. Patients receive docetaxel IV, carboplatin IV, and trastuzumab IV over 30 minutes on day 1 in course 2-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: docetaxel
- Arm II (Experimental): Patients receive oral lapatinib ditosylate once daily on days 1-21 in course 1. Patients receive docetaxel IV and carboplatin IV on day 1 and oral lapatinib ditosylate once daily on days 1-21 in courses 2-7.Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: docetaxel; Drug: lapatinib ditosylate
- Arm III (Experimental): Patients receive trastuzumab IV over 90 minutes on day 1 and oral lapatinib ditosylate daily on days 1-21. Starting on day 22, patients receive docetaxel IV, carboplatin IV, and trastuzumab IV three times a week and oral lapatinib ditosylate once daily on days 1-21 in courses 2-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: docetaxel; Drug: lapatinib ditosylate

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Arms: Arm I; Arm III
Drug: carboplatin — Given IV
Drug: docetaxel — Given IV
Drug: lapatinib ditosylate — Given orally
  Arms: Arm II; Arm III

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether docetaxel and carboplatin are more effective when given together with trastuzumab and/or lapatinib in treating women with stage I, stage II, or stage III breast cancer.

PURPOSE: This randomized phase II trial is studying how well docetaxel and carboplatin work when given together with trastuzumab and/or lapatinib in treating women with stage I, stage II, or stage III breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the clinical efficacy of neoadjuvant docetaxel and carboplatin in combination with trastuzumab (Herceptin®) and/or lapatinib ditosylate by estimating the pathologic complete response (pCR) rate in the breast and axilla of women with HER2/neu-positive resectable stage I-III adenocarcinoma of the breast.

Secondary

* To estimate the molecular effects of lapatinib ditosylate and trastuzumab alone or in combination on tumor tissues of these patients by assessing changes in gene expression using serial gene microarray analysis.
* To assess for gene expression and/or biomarker changes that may be correlated with or predict pCR and clinical response to lapatinib ditosylate and/or trastuzumab in these patients.
* To evaluate the safety and tolerability of these regimens in these patients.
* To evaluate the clinical efficacy of these regimens by estimating the clinical objective response rate (complete response and partial response) in these patients.
* To estimate the rate of congestive heart failure or drop in LVEF (> 10% points from baseline and below lower limits of normal) in each of the three treatment arms.

OUTLINE: This is a multicenter study. Patients are stratified according to baseline tumor size (≤ 3 cm vs > 3 cm) and hormone receptor status (estrogen receptor [ER]- and/or progesterone receptor [PR]-positive vs ER- and PR- negative). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive a trastuzumab IV over 90 minutes on day 1 in course 1. Patients receive docetaxel IV, carboplatin IV, and trastuzumab IV over 30 minutes on day 1 in courses 2-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral lapatinib ditosylate once daily on days 1-21 in course 1. Patients receive docetaxel IV, carboplatin IV as in arm I and oral lapatinib ditosylate once daily on days 1-21 in courses 2-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive trastuzumab IV as in arm I on day 1 and oral lapatinib ditosylate as in arm II on days 1-21 in course 1. Patients receive docetaxel IV, carboplatin IV, and trastuzumab IV as in arm I on day 1 and oral lapatinib ditosylate as in arm II on days 1-21 in courses 2-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Within 4-6 weeks after completion of chemotherapy, all patients under go definitive surgery and/or radiotherapy at the discretion of the treating physician. Tumor biopsy and blood samples are collected for biomarker analysis and molecular analysis at baseline, after course 1, and at the time of definitive breast surgery or completion of chemotherapy. Gene expression changes are analyzed by mRNA microarray analysis and molecular changes in protein expression profiles by IHC. Samples may also be analyzed by RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 70 years, inclusive
* Histologically or cytologically confirmed adenocarcinoma of the breast
* Stage I, II or III disease (early stage) with tumor measuring ≥ 1 cm and meeting any the following criteria:

  * Grade > 1
  * Estrogen receptor- and progesterone receptor-negative
  * Age ≤ 35 years
* HER2/neu-positivity by fluorescence in situ hybridization (FISH)
* Estrogen and progesterone receptor status known prior to study entry.
* ECOG performance status 0-1 Adequate organ function (ejection fraction>- lower limit of normal) as determined by MUGA or echocardiogram.
* If female of childbearing potential, pregnancy test is negative and is willing to use effective contraception while on treatment and for at least 3 months after the last dose of study therapy.
* patient is accessible and willing to comply with treatment, tissue acquisition and follow up.
* patient is willing to provide written informed consent prior to performance of any study-related procedure.
* Adequate organ function as defined by the following laboratory values
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine < 1.5 mg/dL
* Total bilirubin ≤ 1.0 times upper limit of normal (ULN) (< 3 times ULN in patients with Gilbert's syndrome confirmed by genotyping or Invader UGTIA1 molecular assay)
* Alkaline phosphatase (AP), ALT, and AST must meet 1 of the following criteria:
* AP normal AND AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* AP ≤ 2.5 times ULN AND ALT/AST ≤ 1.5 times ULN
* AP ≤ 5 times ULN AND AST/ALT normal

Exclusion Criteria:

* Inflammatory breast cancer, defined as the presence of erythema or induration involving > 1/3 of the breast
* Bilateral invasive breast cancer
* Metastatic disease
* Concurrent therapy with any other non-protocol anti-cancer therapy
* history of any other malignancy within the past 5 years, with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix
* pre-existing motor or sensory neurotoxicity ≥ grade 2 by NCI NTCAE version 3.0
* cardiac disease including any of the following:
* Myocardial infarction within the past 6 months
* Unstable angina
* New York Heart Association class II-IV congestive heart failure
* inflammatory bowel disease or other bowel condition causing chronic diarrhea and requiring active therapy
* active, uncontrolled infection requiring parenteral antimicrobials
* known hypersensitivity to Chinese hamster ovary products or other recombinant human or humanized antibodies and/or known hypersensitivity to any of the study drugs or their ingredients (e.g., polysorbate 80 in docetaxel)
* other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of study drugs or place the subject at undue risk for treatment complications
* hormonal agent (e.g., raloxifene, tamoxifen citrate, or other selective estrogen receptor modulators) for osteoporosis or prevention of breast cancer. subjects must have discontinued these agents 14 days prior to first baseline biopsy.
* prior ipsilateral radiotherapy for invasive or noninvasive breast cancer or to the ipsilateral chest wall for any malignancy
* prior chemotherapy, radiotherapy, or endocrine therapy for currently diagnosed invasive or noninvasive breast cancer
* concurrent ovarian hormonal replacement therapy. Prior treatment must be stopped prior to first baseline biopsy.
* male subjects
* pregnant or lactating subjects

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 7 months

SECONDARY OUTCOMES:
Comparison of pCR rates | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (15):
- United States (15):
  - Central Hematology Oncology Medical Group, Incorporated - Alhambra, Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Jude Heritage Medical Group at Virginia K. Crosson Cancer Center, Fullerton, California
  - North Valley Hematology-Oncology Medical Group, Northridge, California
  - Wilshire Oncology Medical Group, Incorporated - Pomona, Pomona, California
  - Sansum Medical Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Santa Barbara Hematology Oncology - Solvang, Solvang, California
  - Cancer Care Associates Medical Group, Incorporated - Redondo Beach, Torrance, California
  - Cancer Institute of Florida, PA - Orlando, Orlando, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Hematology and Oncology Consultants, PA - Orlando, Orlando, Florida
  - Providence Medical Group, Haute Terre, Indiana
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - New Mexico Cancer Center, Albuquerque, New Mexico

REFERENCES:
- [Derived] Hurvitz SA, Caswell-Jin JL, McNamara KL, Zoeller JJ, Bean GR, Dichmann R, Perez A, Patel R, Zehngebot L, Allen H, Bosserman L, DiCarlo B, Kennedy A, Giuliano A, Calfa C, Molthrop D, Mani A, Chen HW, Dering J, Adams B, Kotler E, Press MF, Brugge JS, Curtis C, Slamon DJ. Pathologic and molecular responses to neoadjuvant trastuzumab and/or lapatinib from a phase II randomized trial in HER2-positive breast cancer (TRIO-US B07). Nat Commun. 2020 Nov 17;11(1):5824. doi: 10.1038/s41467-020-19494-2. PMID 33203854